CLINICAL TRIAL: NCT03960346
Title: Cryoballoon Pulmonary Vein Isolation and Associated Esophageal Effects (Medtronic EGD)
Brief Title: Cryoballoon and Associated Esophageal Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 015-238
Record Dates: First submitted 2016-03-25; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2018-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Esophageal Effects (Other): To determine the correlation between rate of temperature decline and nadir cryoballoon temperatures rate of temperature decline and nadir esophageal temperatures during pulmonary vein isolation. Esophageal temperature probe is used during cryoablation to measure temperatures and then a 4-7 days post procedure esophagoscopy is performed to evaluate the physical effects on the esophagus.
  Interventions: Procedure: Ablation with cryoenergy

INTERVENTIONS:
Procedure: Ablation with cryoenergy — Esophageal temperature-guided ablation using cryoengery and an esophageal temperature probe.
  Other Names: esophageal temperature-guided ablation

SUMMARY:
The primary objectives are to determine the correlation between rate of temperature decline and nadir cryoballoon temperatures rate of temperature decline and nadir esophageal temperatures during pulmonary vein isolation. To accurately measure the distance between the esophagus and the ostium of each pulmonary vein intra-operatively. To attempt to create recommendations for esophageal temperature-guided ablation in order to increase the safety profile of cryoballoon pulmonary vein isolation (PVI) by providing one center's experience. By trending cryoballoon ablation temperatures and subsequent esophageal temperatures, data trends may emerge and be predictive for esophageal ulceration formation. These trends may include:

* Distance between esophagus and pulmonary vein in patients who developed post-ablation esophageal ulcerations
* Intra-procedure esophageal temperatures in patients who developed post-ablation esophageal ulcerations
* Intra-procedure cryoballoon temperatures in patients who developed post-ablation esophageal ulcerations As well as to associate the development of symptoms (including dysphagia, chest pain, fever, "heartburn," or odynophagia) with the presence of ulcerations.

DETAILED DESCRIPTION:
When treating atrial fibrillation and targeting various areas in the left atrium, electrophysiologists have the choice to perform ablation with RF energy or cryoenergy. Esophageal ulceration and in more rare cases, esophageal fistulae, are known complications of this ablation procedure. Though rare (0.1-0.25% fistula rate and 15-20% esophageal ulceration rate according to the most recent Heart Rhythm Society EHRA ECA consensus statement)1, the investigators would very much like to understand how to completely prevent these occurrences. Cryoenergy has more recently been introduced as an energy source used in the PVI procedure; therefore, for this energy source, rates of esophageal ulceration are not yet well-defined. Nine esophageal fistulae have occurred in the first approximately 130,000 cryoballoon procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent, symptomatic, drug-refractory, paroxysmal atrial fibrillation with planned cryoballoon pulmonary vein isolation
2. Age >18 years
3. Planned AF cryoablation procedure

Exclusion Criteria:

1. LA diameter >55mm
2. Severe LVH (LV wall ≥ 15mm)
3. LA thrombus
4. Decompensated heart failure
5. Plans for left atrial ablation lesions beyond isolation of the pulmonary veins
6. History of previous pulmonary vein isolation
7. Inability to place esophageal temperature probe or TEE probe
8. Previously documented phrenic nerve injury
9. Known esophageal pathology (complete GI history worksheet)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-11-25 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Rate of temperature decline | Up to 3 years
  Compare the correlation between rate of temperature decline and nadir cryoballoon temperatures rate of temperature decline and nadir esophageal temperatures during pulmonary vein isolation using a esotest probe esophageal temperature probe to record the esophageal temperatures
Associate the development of symptoms | Up to 3 years
  To associate the development of symptoms (including dysphagia, chest pain, fever, "heartburn," or odynophagia) with the presence of ulcerations using a symptom questionnaire and visualize the esophagus 4-7 days post procedure via esophagoscopy

SECONDARY OUTCOMES:
Phrenic nerve injury | Up to 3 years
  To collect data phrenic nerve injury assessed with patient symptom questionnaire
Post procedure symptoms | Up to 3 years
  To collect data regarding post-procedure symptoms including but not limited to cough, hemoptysis, and pericardial effusion using a symptom questionnaire